CLINICAL TRIAL: NCT01269216
Title: A Randomized Phase II Study of Neoadjuvant Chemoradiotherapy With 5-FU/Leucovorin (FL) vs. TS-1/Irinotecan in Patients With Locally Advanced Rectal Cancer
Brief Title: A Study of Neoadjuvant Chemoradiotherapy With 5-FU/Leucovorin (FL) vs. TS-1/Irinotecan in Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0361
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; titanium silicide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-FU with leucovorin (Active Comparator)
  Interventions: Drug: 5-FU with leucovorin
- TS-1 with Irinotecan (Active Comparator)
  Interventions: Drug: TS-1 with Irinotecan

INTERVENTIONS:
Drug: 5-FU with leucovorin — 5FU 400mg/m2/day with Leucovorin 20mg/m2/day IV on day 1 and day29
  Arms: 5-FU with leucovorin
Drug: TS-1 with Irinotecan — Irinotecan 40mg/m2/day IV on day 1,8,15,22 and 29 with TS-1 70mg/m2/day PO for 25 days
  Arms: TS-1 with Irinotecan

SUMMARY:
This is an open-label, randomized phase II study. Patients will be randomly assigned to either FL or TS-1/irinotecan preoperative chemotherapy regimens by stratification. Patients in FL group will be treated with bolus injections of 5-FU 400 mg/m2/day and LV 20 mg/m2/day for 3 consecutive days every 4 weeks for 2 cycles, and patients in TS-1/irinotecan will be treated with irinotecan 40 mg/m2/day on days 1, 8, 15, 22, 29. TS-1 at a dose of 35mg/m2 was administered orally twice a day after a meal on the day of irradiation (Monday-Friday) concurrent with radiotherapy.

DETAILED DESCRIPTION:
This is an open-label, randomized phase II study. Patients will be randomly assigned to either FL or TS-1/irinotecan preoperative chemotherapy regimens by stratification. Patients in FL group will be treated with bolus injections of 5-FU 400 mg/m2/day and LV 20 mg/m2/day for 3 consecutive days every 4 weeks for 2 cycles, and patients in TS-1/irinotecan will be treated with irinotecan 40 mg/m2/day on days 1, 8, 15, 22, 29. TS-1 at a dose of 35mg/m2 was administered orally twice a day after a meal on the day of irradiation (Monday-Friday) concurrent with radiotherapy. Total 45-50.4 Gy radiations in 25-28 fractions to tumor and draining lymph nodes will be delivered concurrently. Curative surgery (especially total mesorectal excision will be considered as 1st choice of surgical procedure) will be performed for about 4-8 weeks after the completion of chemoradiotherapy. Postoperative chemotherapy regimen is 5-FU plus leucovorin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum
* AJCC/UICC pathologic stages of cT3-4 or cN plus
* Male or female patients, 18 years of age or older
* Be ambulatory and have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* No prior chemotherapy, radiotherapy and immunotherapy
* Adequate major organ functions as following: Hematopoietic function: ANC (absolute neutrophil count)1,500/mm3, Platelet 100,000/mm3, and Hepatic function: serum bilirubin < 1.5 x ULN, AST/ALT levels < 2.5 x ULN, and Renal function: serum creatinine < 1.5 x ULN or Ccr 50 ml/min by Cockcroft formula
* Be willing and able to comply with the protocol for the duration of the study.
* Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Any histologic feature other than adenocarcinoma or arisen from chronic inflammatory bowel disease
* Patients treated with previous surgery, chemotherapy and/or radiotherapy
* Uncontrolled or severe cardiovascular disease: New York Heart Association class III or IV heart disease, and Unstable angina or myocardial infarction within the past 6 months, and History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality.
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
* Other malignancy within the past 5 years except non-melanomatous skin cancer or carcinoma in situ of the cervix.
* Organ allografts requiring immunosuppressive therapy.
* Psychiatric disorder or uncontrolled seizure that would preclude compliance.
* Pregnant, nursing women or patients with reproductive potential without contraception.
* Patients receiving a concomitant treatment with drugs interacting with 5-FU or irinotecan such as flucytosine, phenytoin, or warfarin et al.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Known hypersensitivity to any of the components of the study medications.
* Received any investigational drug or agent within 4 weeks before beginning treatment with study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
pathologic complete response rate | every 4 weeks in FL group, every 2 weeks in TS-1/irinotecan group
  To evaluate pathologic complete response rate in patients with resectable rectal cancer teated with neoadjuvant chemoradiotherapy with 5-FU/leucovorin (FL) vs. TS-1/Irinotecan and surgery followed by fluoropyrimidine based adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea